CLINICAL TRIAL: NCT06106451
Title: Optimization Post-TAVR to IMprove Activity Levels (OPTIMAL Study)
Acronym: OPTIMAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Catalyst Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00324628
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Aortic Valve Disease; Aortic Valve Replacement
Keywords: aortic valve replacement; minimally invasive transcatheter aortic valve replacement; TAVR
MeSH Terms: conditions — Aortic Valve Disease | interventions — Standard of Care; Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to one of the 3 arms of the study.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of Care plus Enhanced Patient Education (Active Comparator): Each participant in this arm will receive enhanced patient education. The research staff will discuss the benefits of cardiac rehabilitation and provide a pamphlet describing the benefits discussed. The research staff will also call the patient four times throughout their participation in the study to encourage physical activity. The enhanced patient education program will begin approximately 2 weeks after the TAVR procedure.
  Interventions: Behavioral: Standard of Care plus Enhanced Patient Education
- Motivational Interviewing Intervention (Active Comparator): Each participant in this arm will have a motivational interviewing program created by a psychologist. The motivational interviewing program will be tailored to the individual participant. The goal of the motivational interviewing program is improved adherence to standard of care cardiac rehabilitation. The motivational interviewing program will begin approximately 2 weeks after the TAVR procedure.
  Interventions: Behavioral: Motivational Interviewing Intervention
- Home-Based Activity Program plus Motivational Interviewing Intervention (Active Comparator): Each participant in this arm will be evaluated by a physical therapist and psychologist. The physical therapist will use the evaluation to create an individually tailored home-based activity program plan. This home-based activity program will be implemented at the 1-month post-operative cardiology clinic appointment. The psychologist will use the evaluation to create an individually tailored motivational interviewing program. The motivational interviewing program will begin approximately 2 weeks after the TAVR procedure.
  Interventions: Behavioral: Home-Based Activity Program plus Motivational Interviewing Intervention

INTERVENTIONS:
Behavioral: Standard of Care plus Enhanced Patient Education — Patients in this arm will receive a pamphlet explaining the benefits of cardiac rehabilitation. This pamphlet will be given in addition to standard of care patient education. The research team will also call the patient at four specified time points to provide additional information.
  Arms: Standard of Care plus Enhanced Patient Education
Behavioral: Motivational Interviewing Intervention — Patients in this arm of the study will participate in a tailor-made motivational interviewing program. These motivational interviewing sessions will focus on enhancing communication with patients. Each motivational interviewing session will be approximately one hour long. There will be a total of 4-6 motivational interviewing sessions.
  Arms: Motivational Interviewing Intervention
Behavioral: Home-Based Activity Program plus Motivational Interviewing Intervention — Patients in this arm will be evaluated on postoperative day 1 by a physical therapist on the study team. After the evaluation, the physical therapist will use the information from the evaluation to make a tailored home-based physical activity program for the patient. The patient will begin the home-based physical activity program on the day of their 1-month post-operative cardiology clinic appointment. In addition to the home-based activity program, patients will participate in a tailor-made motivational interviewing program. These motivational interviewing sessions will focus on enhancing communication with patients. Each motivational interviewing session will be approximately one hour long. There will be a total of 4-6 motivational interviewing sessions.
  Arms: Home-Based Activity Program plus Motivational Interviewing Intervention

SUMMARY:
In this study, the investigators will evaluate the feasibility and potential efficacy of programs to improve functional outcomes after minimally-invasive transcatheter aortic valve replacement (TAVR). The investigators will examine the potential efficacy of (a) a motivation interviewing program, and (b) a home-based physical activity + motivational interviewing program, compared to (c) usual care + enhanced education in patients post-TAVR procedure.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing TAVR procedure
* ≥65 years old
* Ambulatory at baseline without assistance
* Approval of the interventional cardiologist that the patient is an appropriate candidate
* Can access telephone or teleconference

Exclusion Criteria:

* Impaired cognition that would limit participation in study activities
* Medical comorbidities that substantially limit exercise
* Major cardiac comorbidities, including ejection fraction<35%, history of cardiac arrest, complex dysrhythmias at rest, clinically-significant incomplete revascularization, implanted cardiac defibrillator.
* Physical characteristics that substantially limit exercise
* High fall risk (Johns Hopkins Fall Risk Assessment Tool indicating high risk)
* Non-English Speaking
* Vigorous exercise at least 2 times/week for >30 minutes
* Any other physician judgement

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of motivational interviewing sessions attended | Approximately 20 weeks after the day of the TAVR procedure
  This outcome will measure the number of motivational interviewing sessions in which the patient participates. Motivational Interviewing Arm Outcome.
Number of home-based activity sessions attended | Approximately 20 weeks after the day of the TAVR procedure
  This outcome will measure the number of home-based activity sessions the patient logs. Home-based Activity Arm

SECONDARY OUTCOMES:
Number of Cardiac Rehabilitation Sessions Attended | Approximately 20 weeks after the day of the TAVR procedure
  This outcome will measure the number of cardiac rehabilitation sessions attended by the participant.
Number of Barriers to Attending Cardiac Rehabilitation Sessions | Approximately 20 weeks after the day of the TAVR procedure
  This outcome will measure any self-reported barriers that patients experience to participating in cardiac rehabilitation sessions.
Health Status as assessed by the EuroQol 5 Dimension 5 Level (EQ-5D-5L) | Approximately 20 weeks after the day of the TAVR procedure
  This survey is a standardized measure of health status. This survey is scored in two separate sections. The first section measures the five dimensions mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The first section is measured by a minimum score of 5 and a maximum score of 25. Higher score greater level of problems. The second section measures self report health status on a 0 to 100. Higher score best health.
Health Status as assessed by the The Kansas City Cardiomyopathy Questionnaire (KCCQ) | 20 weeks after the day of the TAVR procedure
  The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a survey used to measure health status in patients with heart failure. The KCCQ scores four domains and one summary score. The four domains are physical limitations score, symptom frequency score, quality of life score, and the social limitations score. These five scores are scaled on a scale of 0 to 100. Higher score better health status.
Disability as assessed by the World Health Organization Disability Assessment Schedule (WHO-DAS 2.0) | Approximately 20 weeks after the day of the TAVR procedure
  This survey measures disability due to health conditions including diseases, illnesses, injuries, mental or emotional problems, and problems with alcohol and drugs. This survey has a minimum score of 12 and a maximum score of 60. Higher scores more disability.
Potential Depression as assessed by the Geriatric Depression Scale | 20 weeks after the day of the TAVR procedure
  This survey is a self-reported measure of potential depression in older adults. The minimum score for this survey is 0 and the maximum score is 15. A score of 5 or greater suggests depression.
Safety Events | Approximately 20 weeks after the day of the TAVR procedure
  Any events adverse events or serious adverse events that occur while the patient is participating in the study.
Number of steps as assessed by the 2-Minute Step Test | Approximately 20 weeks after the day of the TAVR procedure
  This test measures the number of steps the patient can take in 2 minutes time. The number of steps recorded is compared to a standardized range of steps based on age.
Number of stands from sitting as assessed by the 30-Second Chair Rise | Approximately 20 weeks after the day of the TAVR procedure
  This test records the number of stands from sitting the patient can complete in 30 seconds time. The number of stands the patient can complete is compared to the average number is compared to the average number in the patient's age group.
The Duration of the Motivational Interviewing Sessions | Approximately 20 weeks after the day of the TAVR procedure
  This outcome will measure the length of each motivational interviewing session attended.
Patient Satisfaction With the Assigned Program | Approximately 20 weeks after the day of the TAVR procedure
  Patient satisfaction will be measured using a Likert scale from 1 to 5. 1 indicates the patient is very dissatisfied. 5 indicates the patient is very satisfied.
Number of Contacts with the Study Physical Therapist | Approximately 20 weeks after the day of the TAVR procedure
  This outcome measure the number of times the patient has contact with the study physical therapy.
Number of steps taken as assessed by Fitbit Data | Approximately 20 weeks after the day of the TAVR procedure
  This outcome will measure activity (e.g. number of steps taken) while wearing the Fitbit.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Brown, MD, Study Director — Johns Hopkins Uiversity; Giancarlo Suffredini, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- The Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
No IPD is anticipated to be shared